CLINICAL TRIAL: NCT00483418
Title: Survey of Testosterone Levels in a Diverse Set of Male Patients With Hormone-Independent Cancers
Brief Title: Survey of Testosterone Levels in Male Cancer Patients
Status: Completed | Type: Observational
Sponsor: Beth Israel Medical Center (Other)
Collaborators: Solvay Pharmaceuticals (Industry); St. Luke's-Roosevelt Hospital Center (Other); Christiana Care Health Services (Other)
Responsible Party: Victoria Rosenwald RN MPH, Beth Israel Oncology Research Office
Other Study IDs: 062-07
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Hypogonadism
Keywords: male; cancer
MeSH Terms: conditions — Hypogonadism; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to survey the total serum testosterone levels in male patients with hormone-independent malignancies. The prevalence of hypogonadism is not known, but is thought to be significant. Results will be adjusted for age and stratified for type of cancer, stage, study site,and presence of opiate use for pain management, which is known to reduce testosterone levels.

DETAILED DESCRIPTION:
Fatigue - extreme tiredness - is associated with cancer as well as its treatment. It has many causes, including the direct effects of the cancer itself, nutritional changes, anemia, changes in activity levels, worry, or, perhaps, hormones such as testosterone. This study is a survey of the amount of testosterone in the blood of men being treated for cancers that are not directly influenced by testosterone (not prostate or testicular tumors).

Testosterone is a hormone that is made by the body from teenage years through adulthood, and helps define male characteristics: sexual function, muscle building, ability to grow hair and deepen the voice. It is believed that the amount of fatigue experienced by men with cancer may be at least and in part due to reduced testosterone levels.

Male cancer patients will be recruited for this study at the time of regularly scheduled visits with their oncologists for treatment or for follow-up care. Patients who agree to participate and sign a consent will be asked to answer questions about their health, medications, vitamins & supplements, and to complete a standardized questionnaire about their quality of life. One tube of blood (8.5 cc) will be drawn at the same time as the other blood tests scheduled for that visit to avoid an additional blood draw. Various elements of the collected information will be compared with the testosterone levels to see if any meaningful patterns exist. The study sample will be drawn from a geographically diverse set of oncology practices in the US. A larger follow-up study is planned if testosterone levels are found to be lower in men with cancer than similar age men without cancer, or if low testosterone levels are associated with more fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Male Cancer patients coming to oncology appointments for treatment or follow-up
* Must be able to answer questionnaire in english, alone or with assistance
* Informed consent

Exclusion Criteria:

* Known HIV infection
* Known hypogonadism
* testosterone or DHEA supplementation within 3 months
* prostate, breast, or testicular cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men with non-hormone dependent cancers who are having blood drawn for other purposes before 12 noon.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart B Fleishman, MD, Principal Investigator — Continuum Cancer Centers of New York
Locations (1):
- Beth Israel Medical Center, New York, New York, United States